CLINICAL TRIAL: NCT01074515
Title: Depression and Functional Outcomes in COPD: Impact of Genetics and Inflammation
Brief Title: Chronic Obstructive Pulmonary Disease (COPD) Activity: Serotonin Transporter (SERT), Cytokines and Depression (CASCADE Study)
Acronym: CASCADE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Collaborators: VA Puget Sound Health Care System (U.S. Federal Agency); The University of Texas Health Science Center at San Antonio (Other); South Texas Veterans Health Care System (U.S. Federal Agency); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Huong Nguyen, Study Principal investigator, University of Washington
Other Study IDs: 37332-B; R01HL093146-01A2 (NIH)
Record Dates: First submitted 2010-02-11; First posted 2010-02-24 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Depression; Inflammation; Genetics; Functioning; Dyspnea; Physical activity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Depression; Inflammation; Dyspnea; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of the study is to look at how genes and certain chemicals in the body are related to depression and chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
Depression is highly prevalent among patients with chronic obstructive pulmonary disease (COPD) and is associated with adverse clinical outcomes. The overall goal of this proposal is to examine the impact of inflammation and genetic risk factors on depression in patients with severe COPD, and to assess the combined effects of inflammation, genetics, and depression on changes in functional outcomes. There is increasing evidence that COPD is associated with systemic inflammation that impacts other organ systems. High levels of systemic inflammatory markers have also been linked to increased risk of depression in both healthy and chronically ill populations. The neurotransmitter serotonin which is involved in the pathophysiology of affective disorders is regulated by the serotonin transporter (SERT) that controls reuptake of serotonin at brain synapses. Recent studies report that SERT polymorphisms are associated with depression, suggesting that variants of this gene may be important in determining whether patients with COPD will develop depression during the course of their disease. The preliminary data linking SERT polymorphisms with depression and data suggesting a relationship between inflammation, depression and COPD strongly argue for a large scale prospective study to critically test these relationships. Therefore, the aims of this prospective study of patients with moderate to very severe COPD are to: 1) Examine the relationship between SERT polymorphisms with depression; 2) Examine the bi-directional longitudinal relationship between markers of systemic inflammation (CRP, IL-1ra, IL-6, IL-12, TNF-α, and IFN-γ) and depressive symptoms in COPD, and explore the role of exacerbations and SERT genotype in this relationship; and 3) Determine the relationship of depression, inflammation, and SERT genotype with decline in functional outcomes (six minute walk test distance, physical activity measured with accelerometers, dyspnea severity, and health related quality of life) in COPD over 2 years. Patients with COPD GOLD Stages II-IV (n=350) will be recruited from two clinical sites over 30 months. Assessments at baseline, year 1 and year 2 will include: blood samples for genotyping (5-HTTLPR, STin2 VNTR, and rs25331) and cytokine assays (CRP, IL-1ra, IL-6, IL-12, TNF-α, and IFN-γ), spirometry, assessment of depression, functional capacity (six minute walk test), performance (physical activity derived from accelerometry), dyspnea, and health related quality of life (HRQL). We will use advanced longitudinal statistical techniques, structural equations modeling and latent growth models, to assess the dynamics of change in depression, inflammation, and functional status as posited by our models as these processes unfold over time.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD confirmed by the following: 1) FEV1/FVC < 70%; 2) Moderate to very severe disease by GOLD criteria (FEV1 <65%); 2) Age > 40 years; and 3) A significant history of current or past cigarette smoking (> 10 pack-years);
* Stable disease with no acute exacerbations of COPD in the past 4 weeks;
* Ability to speak, read and write English

Exclusion Criteria:

* Acute COPD exacerbation within the past 4 weeks (temp exclusion)
* Chronic obstructive lung disorders unrelated to COPD: asthma, bronchiectasis, cystic fibrosis
* Idiopathic Pulmonary Fibrosis
* Congestive Heart Failure
* Chronic renal failure requiring dialysis
* Primary pulmonary vascular disease
* Chronic inflammatory, infectious or auto-immune disease, e.g. osteomyelitis, crohn's disease or rheumatoid arthritis
* Chronic liver disease
* Metastatic cancer
* Chronic antibiotic use or ongoing infection
* Chronic oral prednisone use
* Moderate to severe dementia
* Severe primary mental illness, e.g. schizophrenia, bipolar disease, severe obsessive compulsive disorder
* <2 years life expectancy
* History of fainting with spirometry

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pulmonary and primary care clinics and community sample
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2010-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Depression | 1 year & 2 year

SECONDARY OUTCOMES:
Physical activity by accelerometry | 1 year & 2 year
Dyspnea | 1 year & 2 year
Health related quality of life | 1 year & 2 year
Six Minute Walk Distance | 1 year & 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Huong Q Nguyen, PhD, RN, Principal Investigator — University of Washington; Vincent Fan, MD, MPH, Principal Investigator — Puget Sound Veteran's Affair
Locations (4):
- United States (4):
  - South Texas Veterans Health Care System, San Antonio, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Puget Sound Veterans Administration Health Care System, Seattle, Washington
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Chen Z, Fan VS, Belza B, Pike K, Nguyen HQ. Association between Social Support and Self-Care Behaviors in Adults with Chronic Obstructive Pulmonary Disease. Ann Am Thorac Soc. 2017 Sep;14(9):1419-1427. doi: 10.1513/AnnalsATS.201701-026OC. PMID 28719225
- [Derived] Nguyen HQ, Herting JR, Pike KC, Gharib SA, Matute-Bello G, Borson S, Kohen R, Adams SG, Fan VS. Symptom profiles and inflammatory markers in moderate to severe COPD. BMC Pulm Med. 2016 Dec 3;16(1):173. doi: 10.1186/s12890-016-0330-1. PMID 27914470
- [Derived] Nguyen HQ, Fan VS, Herting J, Lee J, Fu M, Chen Z, Borson S, Kohen R, Matute-Bello G, Pagalilauan G, Adams SG. Patients with COPD with higher levels of anxiety are more physically active. Chest. 2013 Jul;144(1):145-151. doi: 10.1378/chest.12-1873. PMID 23370503